CLINICAL TRIAL: NCT00920972
Title: A Study of Hematopoietic Stem Cell Transplantation (HSCT) in Non-Malignant Disease Using a Reduced-Intensity Preparatory Regime
Brief Title: Campath/Fludarabine/Melphalan Transplant Conditioning for Non-Malignant Diseases
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: St. Louis Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201110144
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Metabolic Disorders; Hematologic, Immune, or Bone Marrow Disorders; Hemoglobinopathies; Non-malignant Disorders
Keywords: Bone marrow; Transplant; Transplantation; Hematopoietic; Umbilical cord; Related; Unrelated; Reduced; Non-myeloablative; Nonmyeloablative; Non-malignant; Nonmalignant
MeSH Terms: conditions — Metabolic Diseases; Hemoglobinopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Stratum 1 (Experimental): Recipients with non-malignant disorders, excluding thalassemia. Related or unrelated 8/8 HLA-matched bone marrow
  Interventions: Drug: Treatment Plan 1: Stratum 1; Drug: GVHD Regimen B: BM Recipients
- Stratum 2 (Experimental): Recipient with transfusion dependent thalassemia. Related or unrelated. 8/8 HLA-matched bone marrow or 5-8/8 HLA-matched UCB
  Interventions: Drug: Treatment Plan 2: Strata 2, 3, or 4; Drug: GVHD Regimen A: UCB Recipients; Drug: GVHD Regimen B: BM Recipients
- Stratum 3 (Experimental): Recipient with hemoglobinopathy Related or unrelated. 7/8 HLA-matched bone marrow or 5-8/8 HLA-matched UCB
  Interventions: Drug: Treatment Plan 2: Strata 2, 3, or 4; Drug: GVHD Regimen A: UCB Recipients; Drug: GVHD Regimen B: BM Recipients
- Stratum 4 (Experimental): Recipient with non-malignant disorder, excluding hemoglobinopathy Related or unrelated. 7/8 HLA-matched bone marrow or 5-8/8 HLA-matched UCB
  Interventions: Drug: Treatment Plan 2: Strata 2, 3, or 4; Drug: GVHD Regimen A: UCB Recipients; Drug: GVHD Regimen B: BM Recipients

INTERVENTIONS:
Drug: Treatment Plan 1: Stratum 1 — Day -50 to -21: Hydroxyurea 30mg/kg PO q day Day -22: Campath-1H 3 mg IV or SQ... Day -21: Campath-1H 10 mg IV or SQ... Day -20: Campath-1H 15 mg IV or SQ... Day -19: Campath-1H 20 mg IV or SQ... Day -8: Fludarabine 30mg/m2 IV... Day -7: Fludarabine 30mg/m2 IV... Day -6: Fludarabine 30mg/m2 IV... Day -5: Fludarabine 30mg/m2 IV... Day -4: Fludarabine 30mg/m2 IV... Day -3: Melphalan 140 mg/m2 IV... (dose modifications for patients <10 kgs) Procedure/Surgery: Hematopoietic stem cell infusion on Day 0...
  Arms: Stratum 1
Drug: Treatment Plan 2: Strata 2, 3, or 4 — Day -50 to -21: Hydroxyurea 30mg/kg PO q day… Day -22: Campath-1H 3 mg IV or SQ... Day -21: Campath-1H 10 mg IV or SQ... Day -20: Campath-1H 15 mg IV or SQ... Day -19: Campath-1H 20 mg IV or SQ... Day -8: Fludarabine 30mg/m2 IV... Day -7: Fludarabine 30mg/m2 IV... Day -6: Fludarabine 30mg/m2 IV... Day -5: Fludarabine 30mg/m2 IV... Day -4: Fludarabine 30mg/m2 IV... Day -4: Thiotepa 8mg/kg IV… Day -3: Melphalan 140 mg/m2 IV... (dose modifications for patients <10 kgs) Procedure/Surgery: Hematopoietic stem cell infusion on day 0...
  Arms: Stratum 2; Stratum 3; Stratum 4
Drug: GVHD Regimen A: UCB Recipients — Day -3: Begin Tacrolimus or cyclosporine Begin MMF Day -1: Abatacept 10mg/kg IV Day +5: Abatacept 10mg/kg IV Day +14: Abatacept 10mg/kg IV Day +28: Abatacept 10mg/kg IV Day +60: Abatacept 10mg/kg IV Day +100: Abatacept 10mg/kg IV
  Arms: Stratum 2; Stratum 3; Stratum 4
Drug: GVHD Regimen B: BM Recipients — Day -3: Begin Tacrolimus or cyclosporine Begin MMF Day -1: Abatacept 10mg/kg IV Day +1: Methotrexate 7.5mg/m2 IV Day +3: Methotrexate 7.5mg/m2 IV Day +5: Abatacept 10mg/kg IV Day +6: Methotrexate 7.5mg/m2 IV Day +14: Abatacept 10mg/kg IV Day +28: Abatacept 10mg/kg IV Day +60: Abatacept 10mg/kg IV Day +100: Abatacept 10mg/kg IV Day +180: Abatacept 10mg/kg IV Day +270: Abatacept 10mg/kg IV Day +365: Abatacept 10mg/kg IV

SUMMARY:
The hypothesis for this study is that a preparative regimen that maximizes host immunosuppression without myeloablation will be well tolerated and sufficient for engraftment of donor hematopoietic cells. It is also to determine major toxicities from these conditioning regimens, within the first 100 days after transplantation.

DETAILED DESCRIPTION:
The study uses reduced intensity conditioning that is immune suppressive to achieve donor cell engraftment without exposure to radiation or high dose chemotherapy in children with non-malignant disorders. The intent is to minimize early and late regimen related toxicities in the context of a reduced intensity regimen.

In addition to maximizing opportunity for donor cell engraftment, the trial seeks to minimize toxicities associated with transplant such as graft versus host disease and employs GVHD prophylaxis that seeks to decrease rates of acute and chronic GVHD in the setting of matched and mismatched donor stem cell transplants from marrow and cord blood sources.

ELIGIBILITY:
Inclusion Criteria:

Stratum 1: Patient must have non-malignant disorder, excluding thalassemia. Must be receiving a 8/8 HLA-matched bone marrow, related or unrelated Stratum 2: Patient must have thalassemia receiving 8/8 HLA-matched bone marrow or 5-8/8 HLA-matched UCB. Related or unrelated.

Stratum 3: Patient must have a hemoglobinopathy receiving 7/8 HLA-matched bone marrow or 5-8/8 HLA-matched UCB. Related or unrelated.

Stratum 4: Patient must have a non-malignant disorder (excluding hemoglobinopathy) receiving 7/8 HLA-matched bone marrow or 5-8/8 HLA-matched UCB. Related or unrelated.

All strata:

* Recipient age < 21 years
* Lansky/Karnofsky >/= 40
* Adequate pulmonary, renal, liver, and other organ function as defined in protocol
* Negative pregnancy test
* Adequate total nucleated cell or CD34+ dose of product as defined in protocol
* If sickle cell, Hemoglobin S <30%

Exclusion Criteria:

* HIV positive
* Invasive infection
* Pregnancy/lactating

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 220 (Estimated)
Dates: Start 2001-12; Primary Completion 2026-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Donor engraftment as measured by chimerism | 100 days post-transplant
  Engraftment is measured in myeloid and lymphoid lineage cells
Major toxicities as graded by the CTC v4 | 100 days post-transplant
  Toxicity monitoring includes unanticipated side effects (new) and all severe irreversible toxicities Grade 3 and above unexpected Grade 4 and above - all toxicities that are possibly, probably or definitely related to protocol therapy All deaths irrespective of attribution

SECONDARY OUTCOMES:
Time to neutrophil and platelet engraftment as measured by complete blood counts | Post transplant
  Defined as an ANC >500/microliter and platelets >20,000 or 50,000/microliter depending on disorder
Incidence of acute graft-versus-host disease as measured by protocol grading scale | 100 days post-transplant
  aGVHD - involving the skin, gut and liver. Classified according to grading described by Thomas et al. NEJM 1975; 292:895-902
Incidence of chronic graft-versus-host disease as measured by protocol grading scale | 2 years post-transplant
  cGVHD classified per Schulman et al. Am J Med 69: 204-17, 1980.
Long-term donor engraftment by donor chimerism | 2 years post-transplant
  Donor chimerism is determined by PCR analysis after cell separation into lymphoid and myeloid lineage cells using antibodies. Can also be detected by FISH analysis in the event of donor and recipient sex discrepancy.
Immune reconstitution by laboratory evaluations | 1 year post-transplant
  Immune reconstitution detected by absolute numbers of T cell phenotypes, B cells and NK cells. T cell function determined by proliferative response to mitogens. B cell function determined by evaluating anti-tetanus antibody titers.
Overall and disease free survival | 2 years post-transplant
  Overall survival is defined as survival with or without disease Event free survival is defined as disease free, severe GVHD free survival, monitoring quality of life and relevant parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Shenoy, MD, Principal Investigator — Washington University School of Medicine (in St. Louis)
Locations (18):
- United States (17):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital of Orange County, Orange, California
  - University of California, San Diego, California
  - Yale School of Medicine, New Haven, Connecticut
  - George Washington University School of Medicine, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Children's Memorial Hospital, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - St. Louis University, St Louis, Missouri
  - Washington University School of Medicine (in St. Louis), St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Medical Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - The University of Oklahoma, Oklahoma City, Oklahoma
  - Texas Transplant Institute, San Antonio, Texas
- University of Calgary, Calgary, Canada

REFERENCES:
- [Result] Bhatla D, Davies SM, Shenoy S, Harris RE, Crockett M, Shoultz L, Smolarek T, Bleesing J, Hansen M, Jodele S, Jordan M, Filipovich AH, Mehta PA. Reduced-intensity conditioning is effective and safe for transplantation of patients with Shwachman-Diamond syndrome. Bone Marrow Transplant. 2008 Aug;42(3):159-65. doi: 10.1038/bmt.2008.151. Epub 2008 May 26. PMID 18500373
- [Result] Hansen MD, Filipovich AH, Davies SM, Mehta P, Bleesing J, Jodele S, Hayashi R, Barnes Y, Shenoy S. Allogeneic hematopoietic cell transplantation (HCT) in Hurler's syndrome using a reduced intensity preparative regimen. Bone Marrow Transplant. 2008 Feb;41(4):349-53. doi: 10.1038/sj.bmt.1705926. Epub 2007 Nov 19. PMID 18026148
- [Result] Rao A, Kamani N, Filipovich A, Lee SM, Davies SM, Dalal J, Shenoy S. Successful bone marrow transplantation for IPEX syndrome after reduced-intensity conditioning. Blood. 2007 Jan 1;109(1):383-5. doi: 10.1182/blood-2006-05-025072. Epub 2006 Sep 21. PMID 16990602
- [Result] Shenoy S, Grossman WJ, DiPersio J, Yu LC, Wilson D, Barnes YJ, Mohanakumar T, Rao A, Hayashi RJ. A novel reduced-intensity stem cell transplant regimen for nonmalignant disorders. Bone Marrow Transplant. 2005 Feb;35(4):345-52. doi: 10.1038/sj.bmt.1704795. PMID 15592491
- [Derived] King AA, Kamani N, Bunin N, Sahdev I, Brochstein J, Hayashi RJ, Grimley M, Abraham A, Dioguardi J, Chan KW, Douglas D, Adams R, Andreansky M, Anderson E, Gilman A, Chaudhury S, Yu L, Dalal J, Hale G, Cuvelier G, Jain A, Krajewski J, Gillio A, Kasow KA, Delgado D, Hanson E, Murray L, Shenoy S. Successful matched sibling donor marrow transplantation following reduced intensity conditioning in children with hemoglobinopathies. Am J Hematol. 2015 Dec;90(12):1093-8. doi: 10.1002/ajh.24183. Epub 2015 Oct 6. PMID 26348869